CLINICAL TRIAL: NCT05651243
Title: Non-pharmacological Treatments for Obesity: Leveraging the Appetite Suppressive Effects of Hyperketonemia Through Exogenous Ketone Ingestion to Treat Obesity, Insulin Resistance, and Cognition
Brief Title: Ketone Esters for Appetite, Cognition, and Cardiovascular Function in Individuals With Obesity and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Mississippi (Other)
Responsible Party: Principal Investigator, Austin Graybeal, Assistant Professor, University of Southern Mississippi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22-877
Record Dates: First submitted 2022-11-03; First posted 2022-12-14 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone Ester (Experimental): Oral ketone ester supplement
  Interventions: Dietary Supplement: Ketone Ester Supplement
- Placebo (Placebo Comparator): Taste and viscosity matched placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone Ester Supplement — Oral ingestion of a ketone supplement combined with a flavoring agent and diluted in water
  Arms: Ketone Ester
Other: Placebo — Oral ingestion of cellulose combined with a flavoring agent and diluted in water
  Arms: Placebo

SUMMARY:
The goal of this single-blind randomized placebo-controlled trial is to test the effects of an oral ketone supplement on appetite, cognition, metabolism, and cardiovascular function in individuals with obesity and insulin resistance.

The main question[s] it aims to answer are:

* Does taking the ketone supplement reduce appetite and improve cognition?
* How does the ketone supplement alter metabolism and cardiovascular function?

Participants will be asked to consume a randomly assigned ketone ester supplement or a placebo and testing will be done to see how the supplement affects the following compared to a placebo:

* appetite,
* cognition,
* metabolism
* cardiovascular function

Researchers will compare individuals with obesity and insulin resistance to individuals with normal weight and no insulin resistance to see if the ketone supplement affects groups differently.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-50 years of age.
* Presence of metabolic sydnrome

Control Participant Eligibility:

* A waist circumference of < 102 cm for males and < 88 cm for females, and
* No indication of metabolic syndrome

Exclusion Criteria:

* Pregnant
* Breastfeeding or lactating
* Missing any limbs or part of a limb
* Having a substantial amount of metal implants (metal plates or complete joint replacements)
* Having a pacemaker or any other electrical implant
* Type I diabetes
* Gestational diabetes
* Taking insulin
* Any history of severe traumatic brain injury or mild traumatic brain injury within the last two years
* Kidney disease
* Liver disease
* Thyroid disease
* Any diagnosed neurological or neurodegenerative diseases
* Any surgeries that would impact swallowing and/or digestion
* Being on a ketogenic diet or having been on a ketogenic diet in the last 6 months
* Having received ionizing radiation from a medical procedure within the last 30 days
* Being on a medically prescribed diet

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Baseline (pre-ingestion)
  Blood pressure responses (systolic and diastolic) to sympathoexcitation
Blood pressure | 30 minutes post ingestion
  Blood pressure responses (systolic and diastolic) to sympathoexcitation
Blood pressure | 45 minutes post ingestion
  Blood pressure responses (systolic and diastolic) to sympathoexcitation
Blood pressure | 60 minutes post ingestion
  Blood pressure responses (systolic and diastolic) to sympathoexcitation
Blood pressure | 75 minutes post ingestion
  Blood pressure responses (systolic and diastolic) to sympathoexcitation
Blood pressure | 90 minutes post ingestion
  Blood pressure responses (systolic and diastolic) to sympathoexcitation
Blood pressure | 105 minutes post ingestion
  Blood pressure responses (systolic and diastolic) to sympathoexcitation
Heart Rate | Baseline (pre-ingestion)
  Heart rate responses to sympathoexcitation
Heart Rate | 30 minutes post ingestion
  Heart rate responses to sympathoexcitation
Heart Rate | 45 minutes post ingestion
  Heart rate responses to sympathoexcitation
Heart Rate | 60 minutes post ingestion
  Heart rate responses to sympathoexcitation
Heart Rate | 75 minutes post ingestion
  Heart rate responses to sympathoexcitation
Heart Rate | 90 minutes post ingestion
  Heart rate responses to sympathoexcitation
Heart Rate | 105 minutes post ingestion
  Heart rate responses to sympathoexcitation
Heart Rate Variability | Baseline (pre-ingestion)
  Index of cardiac autonomic control
Heart Rate Variability | 45 post ingestion
  Index of cardiac autonomic control
Cardiac Baroreflex Sensitivity | 105 minutes post ingestion
  Changes in cardiac interval relative to changes in systolic blood pressure
Hunger - Visual Digital Analog Scale (0-100) | Baseline, 30, 45, 60, 75, 90, 105, 120 minutes post ingestion
  Changes in subjective rating of hunger
Fullness - Visual Digital Analog Scale (0-100) | Baseline, 30, 45, 60, 75, 90, 105, 120 minutes post ingestion
  Changes in subjective rating of fullness
Desire to eat - Visual Digital Analog Scale (0-100) | Baseline, 30, 45, 60, 75, 90, 105, 120 minutes post ingestion
  Changes in subjective rating of desire to eat
Prospective consumption of food - Visual Digital Analog Scale (0-100) | Baseline, 30, 45, 60, 75, 90, 105, 120 minutes post ingestion
  Changes in subjective rating of prospective consumption of food
Thirst - Visual Digital Analog Scale (0-100) | Baseline, 30, 45, 60, 75, 90, 105, 120 minutes post ingestion
  Changes in subjective rating of thirst
Stroop Test - Digital Cognitive Function Test | Baseline, 75 minutes
  Changes in Stroop score
Go/No-go Test - Digital Cognitive Function Test | Baseline, 75 minutes
  Changes in Go/No-go score
Task Switching Task - Digital Cognitive Function Test | Baseline, 75 minutes
  Changes in Task Switching Task score
Number Back Test - Digital Cognitive Function Test | Baseline, 75 minutes
  Changes in Number Back Test score
Digit Span Test - Digital Cognitive Function Test | Baseline, 75 minutes
  Changes in Digit Span Test score

SECONDARY OUTCOMES:
Prefrontal Cortex Oxygenation | Baseline, 90 minutes post ingestion
  Near-infrared spectroscopy
Peripheral Blood Flow | Baseline, 30, 60 and 90 minutes post ingestion
  Doppler Ultrasound of Femoral Artery
Peripheral Vascular Conductance | Baseline, 30, 60 and 90 minutes post ingestion
  Blood flow normalized to blood pressure (mL/min/mmHg)
Blood ketones | Baseline, 30, 60, 90, 120 minutes post ingestion
  Ketone body level from capillary blood
Blood glucose | Baseline, 30, 60, 90, 120 minutes post ingestion
  Blood glucose level from capillary blood
Oxygen Consumption from Respiratory Gases | Baseline and continuous for 120 minutes
  Amount of oxygen consumed using indirect calorimetry
Carbon Dioxide Produced from Respiratory Gases | Baseline and continuous for 120 minutes
  Amount of carbon dioxide produced using indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Austin J Graybeal, PhD, Principal Investigator — University of Southern Mississippi
Locations (1):
- University of Southern Mississippi - School of Kinesiology and Nutrition, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stavres J, Aultman RS, Brandner CF, Vallecillo-Bustos A, Compton AT, Swafford SH, Newsome TA, Graybeal AJ. Influence of exogenous ketosis on spontaneous cardiovagal baroreflex gain and blood pressure responses to isometric handgrip in individuals with metabolic syndrome: a placebo-controlled pilot study. Eur J Appl Physiol. 2025 Jul 31. doi: 10.1007/s00421-025-05921-z. Online ahead of print. PMID 40745496